CLINICAL TRIAL: NCT03374176
Title: Efficacy of Amoxicillin-metronidazole Compared to Clindamycin in the Treatment of Periodontitis in Patients With Diabetes
Brief Title: Efficacy of Amoxicillin-metronidazole Compared to Clindamycin in Patients With Periodontitis and Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centro Universitario de Tonalá (Other)
Responsible Party: Principal Investigator, Arieh Roldán Mercado Sesma, Research professor associate B, Centro Universitario de Tonalá
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CUT2017002
Record Dates: First submitted 2017-12-12; First posted 2017-12-15 (Actual); Results first posted 2020-06-23 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Periodontitis; Periodontal Pocket; Diabetes Mellitus
Keywords: periodontitis; diabetes mellitus; systemic antimicrobials
MeSH Terms: conditions — Periodontitis; Periodontal Pocket; Diabetes Mellitus | interventions — Amoxicillin; Metronidazole; Clindamycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AMX-MET (Active Comparator): AMX-MET Amoxicillin 500 mg + Metronidazole 250 mg. Capsules.
  1 capsule tid during 7 days.
  Interventions: Drug: Amoxicillin 500 mg / Metronidazole 250 mg
- Clindamycin (Experimental): Clindamycin Clindamycin 300 mg + placebo. Capsules.
  1 capsule tid during 7 days.
  Interventions: Drug: Clindamycin 300 mg

INTERVENTIONS:
Drug: Amoxicillin 500 mg / Metronidazole 250 mg — Subjects were instructed to take a capsule three times a day for 7 days
  Arms: AMX-MET
Drug: Clindamycin 300 mg — Subjects were instructed to take a capsule three times a day for 7 days
  Arms: Clindamycin

SUMMARY:
Periodontitis is an inﬂammation of the supporting structures of the teeth, usually caused by speciﬁc or groups of microorganisms that results in the progressive destruction of the periodontal ligament and alveolar bone. the objective of periodontitis treatment is to reduce the number of periodontal pathogens. However, there is not an agreement in the use of systemic antibiotics in patients with diabetes. The purpose of the present study was to determine the efficacy of amoxicillin/metronidazole compared to clindamycin during non-surgical treatment of periodontitis in patients with type 2 diabetes mellitus.

Patients and methods In this double-blind, randomized clinical trial, a total of 42 patients with chronic periodontitis and type 2 diabetes were included in a 24-months follow-up. Patients were randomly assigned to treatment with either amoxicillin/metronidazole or clindamycin every for 7 days. Clinical determinations (depth of probing, bleeding at the probe and plaque index) were performed to determine the extent and severity of periodontitis before and after the pharmacological treatment. The intra-group differences were calculated with Wilcoxon rank test. The inter-group differences were calculated with Mann-Whitney test. Sex, bacterial plaque, and bleed to the sounding were summarized using proportions and analyzed with the chi-square method. In all analyses, a P-value of <0.05 (two tailed) was considered statistically significant

DETAILED DESCRIPTION:
A parallel, randomized, double-blind, active controlled, single center clinical trial was designed to compare the efficacy of two antibiotic therapies with 24-month follow-up. The study protocol was approved by the ethical committee of the Universitary Center of Health Sciences of University of Guadalajara and conducted according to Good Clinical Practice and the principles of the Declaration of Helsinki. All patients provided written informed consent before the initiation of study procedures.

A total of 5 non-study subjects with chronic periodontitis were recruited and used for the calibration exercise. Two designated examiners measured full-mouth probing pockets depths (PPD) for all 5 subjects. On the same day (with a minimum of 15 min separation), the examiner repeated the examination. Upon completion of all measurements, the intra-examiner repeatability for PPD measurement was assessed. The examiner was judged to be reproducible after fulﬁlling the pre-determined success criteria (the percentage of agreement within 2 mm between repeated measurements had to be at least 70 %). The examiner showed 78.3 % reproducibility.

The sample size was calculated with a 95% confidence level and statistical power of 80 %. A standard deviation of 1.0 mm with an expected difference of 1.0 mm probing pocket depth reduction between treatments. This resulted in a total of 14 patients per arm, however this sample was increased 20% (21 patients per group) to compensate for possible dropouts.

Patient population Criteria for selection Patients of both sexes (aged >18 to 70 years) with a diagnosis of chronic periodontitis according to the 1999 International World Workshop for a Classification of Periodontal Diseases and Conditions and a history of type 2 diabetes with a HbA1C < 8 % and a fasting plasma glucose (FPG) < 180 mg/dL. Patients with aggressive periodontitis, pregnant or lactating females, required antibiotic pre-medication for the performance of periodontal examination and treatment or received antibiotic treatment in the previous 3 months were excluded. A history of anti-inﬂammatory therapy within preceding six months or that had received a course of periodontal treatment within the last 6 months, allergies to penicillin, metronidazole or clindamycin, and were not able to provide consent to participate in the study were also criteria for exclusion.

Intervention Subjects were randomly allocated 1:1 to receive 500 mg amoxicillin + 250 mg metronidazole or 300 mg clindamycin + placebo using a computer that generated a list of random numbers. Subjects were instructed to take the treatment three times a day for 7 days in both groups.

Assessments During these sessions, a case presentation was given to each subject related to the speciﬁc features of his/her disease, as well as a supra- and sub-gingival mechanical debridement was performed. A complete periodontal examination was performed, including a full medical and dental history, an intra-oral examination and a full-mouth periodontal probing. A radiographic examination was undertaken using either periapical x-rays or a ortopantomography.

Clinical parameters Clinical parameters were assessed using a North Caroline Periodontal Probe by the calibrated examiner at six sites. Full-mouth plaque scores were recorded by assigning a binary score to each surface (1 for plaque present, 0 for absent) and by calculating the percentage of total tooth surfaces that revealed the presence of plaque detected by the use of tablet. Similarly, a full-mouth percentage bleeding score was calculated after assessing dichotomously the presence of bleeding on probing from the bottom of the pocket when probing with a manual probe with a force of 0.3n. Full-mouth PPD and recession of the gingival margin were recorded at the same time with measurements rounded to the nearest millimeter.

Non-surgical periodontal therapy Periodontal therapy was initiated within 1 month of the baseline screening examination. A standard cycle of periodontal therapy consisting of oral hygiene instructions, supra- and sub-gingival mechanical instrumentation of the root surface (scaling and root planning) was performed by two experienced therapists.

Local anesthesia was used as necessary. Patients relied on standard oral hygiene methods as instructed at the commencement of the study.

Post-treatment controls The objectives of the post-treatment appointments were to control and reinforce the oral hygiene habits of each subject, to monitor the early healing events and to report any adverse events or additional medications taken. In addition, the 1-week post-treatment visit served as a compliance control, as subjects were asked to return any medication not taken and/or the empty bottles. The number of pills not taken by the study subjects was documented.

Re-assessment examinations Reassessment visits occurred within a month and a half of the completion of the pharmacological treatment. During these appointments, the examiner recorded any changes in the medical history and repeated clinical periodontal parameters recorded at the basal visit.

Statistical analysis Age, FPG, HbA1C, tooth, and sounding depth were presented in means and standard deviation. The intra-group differences were calculated with Wilcoxon rank test. The inter-group differences were calculated with Mann-Whitney test. Sex, bacterial plaque, and bleed to the sounding were summarized using proportions and analyzed with the chi-square method. In all analyses, a P-value of <0.05 (two tailed) was considered statistically significant. All statistical analyses were conducted using SPSS software (IBM Corporation, Armonk, NY, USA) version 21.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes
* Age >18 to 70 years
* Diagnosis of chronic periodontitis according to the 1999 International World Workshop for a Classification of Periodontal Diseases and Conditions
* History of type 2 diabetes
* HbA1C < 8 %
* Fasting plasma glucose (FPG) < 180 mg/dL.

Exclusion Criteria:

* Aggressive periodontitis
* Pregnant or lactating females,
* Required antibiotic pre-medication for the performance of periodontal examination and treatment or received antibiotic treatment in the previous 3 months were excluded.
* A history of anti-inﬂammatory therapy within preceding six months
* Had received a course of periodontal treatment within the last 6 months,
* Allergies to penicillin, metronidazole or clindamycin,
* Not able to provide consent to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-09 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was carried out on patients at the Integral Dentistry Clinics of the University Center of Health Sciences of the University of Guadalajara in Jalisco, Mexico. The participants attended for dental care from August 2015 to December 2016.
Pre-assignment Details: A radiographic examination was undertaken using either periapical films or a pantomogram. Periodontal therapy was initiated within 1month of the baseline screening examination.
Groups:
- AMX-MET: AMX-MET Amoxicillin 500 mg + Metronidazole 250 mg. Capsules.
  1 capsule tid during 7 days.
  Amoxicillin 500 mg / Metronidazole 250 mg: Subjects were instructed to take a capsule three times a day for 7 days
- Clindamycin: Clindamycin Clindamycin 300 mg + placebo. Capsules.
  1 capsule tid during 7 days.
  Clindamycin 300 mg: Subjects were instructed to take a capsule three times a day for 7 days
Period: Overall Study
Arm/Group | AMX-MET | Clindamycin
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- AMX-MET: 500 mg amoxicillin plus 250 mg metronidazole three times a day for 7days
- Clindamycin: 300mg clindamycin plus placebo three times a day for 7days
- Total: Total of all reporting groups
Arm/Group | AMX-MET | Clindamycin | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (8.0) | 52.0 (10.6) | 52.2 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 11 | 7 | 18
Fasting Plasma Glucose [Mean (Standard Deviation); unit: mg/dL] | 134.1 (23.3) | 136.3 (25.7) | 135.2 (24.2)
HbA1C [Mean (Standard Deviation); unit: %] — HbA1C is reported as a percentage
  % | 7.1 (0.4) | 7.3 (0.4) | 7.2 (0.4)
Number of Teeth present in the subjects [Mean (Standard Deviation); unit: Teeth] | 25 (3) | 24 (5) | 24 (4)
Probing depth [Mean (Standard Deviation); unit: mm] | 2.4 (0.6) | 2.6 (0.6) | 2.5 (0.6)
Sites with Plaque [Mean (Standard Deviation); unit: Sites] — Plaque accumulation:
  0: no plaque
  1. separate flecks of plaque at the cervical margin of the tooth
  2. a thin continuous band of plaque (up to 1 mm) at the cervical margin of the tooth
  3. a continuous band of plaque wider than 1 mm but covering less than one-third of the crown of the tooth
  4. plaque covering at least one-third but less than two-thirds of the crown of the tooth
  5. plaque covering two-thirds or more of the crown of the tooth. Once you have all measures you should calculate a mean of all teeth. The greater index the worse gingival disease.
  Sites | 40.4 (22.9) | 40.7 (21.9) | 40.5 (22.1)
Bleeding on Probing [Mean (Standard Deviation); unit: Sites] — 0: absence of inflammation
  1. mild inflammation; a slight change in color, little change in the texture of any portion of but not the entire marginal or papillary gingival unit
  2. mild inflammation; criteria as above but involving the entire marginal or papillary gingival unit
  3. moderate inflammation; glazing, redness, edema, and/or hypertrophy of the marginal or papillary gingival unit 4; severe inflammation; marked redness, edema, and/or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration.
  The greater index the worse gingival disease
  Sites | 42.4 (24.2) | 55.6 (25.8) | 49.0 (25.6)

OUTCOME MEASURES:

1. Primary Outcome: Probing Depth
Description: The size of the periodontal pocket
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | AMX-MET | Clindamycin
Number analyzed (Participants) | 21 | 21
mm | 0.44 (0.27) | 0.50 (0.17)
Statistical Analysis 1: Comparison: AMX-MET vs Clindamycin; Test type: Equivalence; p < 0.05, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 0.05, Standard Deviation 1; chi-square

2. Secondary Outcome: Sites With Plaques
Description: 0: no plaque
  1. separate flecks of plaque at the cervical margin of the tooth
  2. a thin continuous band of plaque (up to 1 mm) at the cervical margin of the tooth
  3. a continuous band of plaque wider than 1 mm but covering less than one-third of the crown of the tooth
  4. plaque covering at least one-third but less than two-thirds of the crown of the tooth
  5. plaque covering two-thirds or more of the crown of the tooth. A higher scores mean a worse outcome
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: Sites
Arm/Group | AMX-MET | Clindamycin
Number analyzed (Participants) | 21 | 21
Sites | 17.6 (13.3) | 15.8 (10.0)

3. Secondary Outcome: Sites With Bleeding on Probing
Description: Refers to bleeding on probing 0: absence of inflammation
  1. mild inflammation; a slight change in color, little change in the texture of any portion of but not the entire marginal or papillary gingival unit
  2. mild inflammation; criteria as above but involving the entire marginal or papillary gingival unit
  3. moderate inflammation; glazing, redness, edema, and/or hypertrophy of the marginal or papillary gingival unit 4; severe inflammation; marked redness, edema, and/or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: Sites
Arm/Group | AMX-MET | Clindamycin
Number analyzed (Participants) | 21 | 21
Sites | 16.1 (11.2) | 22.1 (12.9)

4. Secondary Outcome: Total Count of All Teeth Lost Across All Participants
Description: The total count of all teeth lost in all participants.
Time Frame: 2 years
Measure: Number; unit: total count of all teeth lost
Arm/Group | AMX-MET | Clindamycin
Number analyzed (Participants) | 21 | 21
total count of all teeth lost | 0 | 0

ADVERSE EVENTS:
Time Frame: The adverse events were collected for 10 days. Seven days during the intervention period and 3 days after the final visit.
Description: No serious adverse events occurred. The definition of adverse event and the serious adverse event is the same from the clinicaltrials.gov
Arm/Group | AMX-MET | Clindamycin
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

LIMITATIONS AND CAVEATS:
The prin- cipal limitation of the present study was the absence of a group with SRP plus placebo. This study design, using a placebo group, could help us to evaluate the efficacy of clindamycin versus SRP alone.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes